CLINICAL TRIAL: NCT07369986
Title: A Phase 2b, Open-Label Study of Iparomlimab and Tuvonralimab to Facilitate Surgery Avoidance in Women With Resectable, Mismatch Repair-Deficient Endometrial Cancer
Brief Title: Immunotherapy for Surgery Avoidance in Vulnerable dMMR Endometrial Cancer
Acronym: IMMUNE-SAVE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2025-811
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Immunotherapy; Mismatch Repair Deficiency
MeSH Terms: conditions — Endometrial Neoplasms; Turcot syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — Iparomlimab and Tuvonralimab as a strategy to facilitate non-surgical management in women with surgically completely resectable dMMR endometrial cancer.

SUMMARY:
Efficacy evaluate of iparomlimab and tuvonralimab (a PD-1/CTLA-4 bispecific antibody) in patients with surgically resectable dMMR endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 years or older.
2. Histologically confirmed endometrial cancer (excluding carcinosarcoma).
3. FIGO (2009) stage I to IIIC2 disease that is considered surgically completely resectable.

Confirmed dMMR or MSI-H, defined by either loss of expression of one or more mismatch repair proteins (MLH1, PMS2, MSH2, MSH6 or MSI-H) for by immunohistochemistry, or MSI-H status confirmed by polymerase chain reaction assay.

5)No prior systemic anti-tumor therapy (including chemotherapy, radiotherapy, targeted therapy, or immunotherapy) within the past 5 years.

6)Eastern Cooperative Oncology Group Performance Status of 0 or 1. 7)Laboratory test results within 7 days prior to the first dose must meet the following criteria. Laboratory values are not valid if the patient received granulocyte colony-stimulating factor or a blood transfusion within 14 days prior to sample collection.

White blood cell count ≥2,000/mm3 and absolute neutrophil count ≥1,500/mm3. Platelet count ≥100,000/mm3. Hemoglobin ≥9.0 g/dL.

Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0-fold of the upper limit of normal (ULN) (or ≤5.0-fold the ULN of the study site in patients with liver metastases). Total bilirubin ≤1.5-fold of the ULN.

Creatinine ≤1.5-fold of the ULN or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) ≥ 45 mL/min.

8)Women of childbearing potential:

* Must agree to use contraception from the time of informed consent until at least 5 months after the last dose of the investigational product.
* Must agree not to breastfeed from the time of informed consent until at least 5 months after the last dose.

Exclusion Criteria:

1)Multiple primary malignancies, except for: adequately resected basal cell or squamous cell carcinoma of the skin (Stage I), superficial bladder cancer, or any other malignancy that has been disease-free for over 5 years.

History of severe hypersensitivity to any monoclonal antibody. 3)Known hypersensitivity to iparomlimab and tuvonralimab or any of their excipients.

4)Concurrent or history of clinically significant autoimmune disease. 5)Current or prior interstitial lung disease or pulmonary fibrosis documented by imaging or clinical assessment. Patients with radiation pneumonitis may be enrolled if it is confirmed to be stable (beyond the acute phase) and without anticipated recurrence.

6)Concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease. 7)Symptomatic pericardial effusion, pleural effusion, or ascites requiring treatment.

8)Uncontrolled tumor-related pain. 9)Transient ischemic attack, cerebrovascular accident, or thromboembolism within 180 days prior to enrollment.

10)Uncontrolled or clinically significant cardiovascular disease, defined as any of the following within 180 days prior to enrollment:

* Myocardial infarction;
* Unstable angina pectoris;
* Congestive heart failure of New York Heart Association (NYHA) Class III or IV
* Poorly controlled hypertension despite appropriate treatment (e.g., sustained systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg for ≥ 24 hours)
* Arrhythmia requiring treatment 11)Requirement for ongoing therapeutic anticoagulation (low-dose aspirin or other antiplatelet therapy is permitted).

  12)Poorly controlled diabetes mellitus. 13)Active systemic infection requiring treatment. Systemic corticosteroid therapy (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before enrollment.

  15)Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular targeted therapy agents, or immunotherapy agents) within 28 days before randomization.

  16)Surgical pleurodesis or pericardium within 28 days prior to enrollment. 17)Major surgery within 4 weeks or minor surgery within 7 days before the first dose, without full recovery. Patients scheduled for major surgery during the study period are excluded (video-assisted thoracoscopic surgery or diagnostic procedures are not considered exclusions if recovery is adequate).

  18)Administration of any therapeutic radiopharmaceutical within 56 days prior to enrollment (diagnostic use is permitted).

  19)Active tuberculosis. 20)Positive serology for human immunodeficiency virus (HIV-1/2 antibody), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody. Patients who are HBsAg-positive may be enrolled if hepatitis B virus DNA is below the lower limit of detection.

  21)Any other severe medical or psychiatric condition, or abnormal laboratory findings, that in the investigator's judgment would increase the risk of study participation, compromise protocol compliance, or interfere with the interpretation of study results.

  22)Participation in another clinical trial and receipt of an investigational product within 4 weeks prior to the first dose.

  23)Pregnancy, lactation, or intention to become pregnant during the study period.

  24)Positive urine pregnancy test within 72 hours before treatment initiation (if urine test is positive or indeterminate, a confirmatory serum pregnancy test is required).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological or clinical complete response rate | From the time of enrollment until 12 months after the completion of treatment

IPD SHARING:
Plan to Share IPD: No